CLINICAL TRIAL: NCT04521842
Title: Influence of Large Head vs Standard Size During Total Hip Arthroplasty on Gait Analysis - Prospective Randomized Controlled Trial
Brief Title: Influence of Femoral Head Size During Total Hip Arthroplasty on Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WarsawMU/Head
Record Dates: First submitted 2020-08-10; First posted 2020-08-21 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis, Hip; Hip Arthritis; Gait, Frontal
Keywords: osteoarthritis; hip; gait; walk; biomechanics
MeSH Terms: conditions — Osteoarthritis, Hip; Gait Disorders, Neurologic; Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Patients qualified to undergo total hip arthroplasty due to the end-stage osteoarthritis will be randomly allocated to receive either standard femoral head size implants nor large ones. Pre- and postoperatively they will undergo gait analysis. To avoid risk of bias assessor will be blinded in terms of used implants in every participants case.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard size femoral head implant (Placebo Comparator): Participants qualified to undergo total hip replacement who will receive standard femoral head size implant
  Interventions: Procedure: Total hip replacement
- Large size femoral head (Active Comparator): Participants qualified to undergo total hip replacement who will receive large femoral head size implant
  Interventions: Procedure: Total hip replacement

INTERVENTIONS:
Procedure: Total hip replacement — Total hip replacement in treatment of end-stage osteoarthritis

SUMMARY:
Total hip replacement (THR) is being considered as one of the most effective medical procedures. Since its introduction, there was a worldwide debate over proper implant selection in terms of size, bearing type and shape. The diameter of used femoral heads components grew throughout the years - from 22 mm in the 1960s to 32 mm in the 2000s, which is the most commonly used size nowadays. In recent years there was a visible use of large femoral heads (>=36mm) in several registers. In the USA there was a significant grow in use of this heads rising from 1% in early 200s to even 58% in 2009. There is a strong evidence data and many researchers concerning range of movement, risk of dislocation, functional results, pain and prosthesis wear depending of femoral head size.

In terms of gait characteristics there are several deviations reported concerning both patients with hip osteoarthritis (OA) and following THR. There is a lack of literature concerning influence of used implants on gait parameters and whether this goal of the surgery can be achieved.

The aim of this study was to assess potential differences of lower limb biomechanics during gait in patients following total hip replacement surgery depending on femoral head diameter and compare them to the normal gait of healthy volunteers. As a secondary outcome authors wanted to inspect correlation between gait parameters and patient-reported outcome.

DETAILED DESCRIPTION:
Total hip replacement (THR) is being considered as one of the most effective medical procedures. Since its introduction, there was a worldwide debate over proper implant selection in terms of size, bearing type and shape. The diameter of used femoral heads components grew throughout the years - from 22 mm in the 1960s to 32 mm in the 2000s, which is the most commonly used size nowadays. In recent years there was a visible use of large femoral heads (>=36mm) in several registers. In the USA there was a significant grow in use of this heads rising from 1% in early 200s to even 58% in 2009. There is a strong evidence data and many researchers concerning range of movement, risk of dislocation, functional results, pain and prosthesis wear depending of femoral head size.

In terms of gait characteristics there are several deviations reported concerning both patients with hip osteoarthritis (OA) and following THR. It is well-proven that those with hip OA have reduced stride length and reduced cadence, reduced gait velocity, and reduced joint excursion. Patients after THR walk with lower hip-abduction moments, sagittal-plane range of motion. It is believed that it might be a consequence of pain-avoidance mechanism developed as an adaptation for joint disease, which is still present after the surgery. What is more, there are publications, which underline that lower limb biomechanics during gait do not return to normal following THR.

However there is a lack of literature concerning influence of used implants on gait parameters and whether this goal of the surgery can be achieved.

According to authors best knowledge this study is the first to ever describe potential differences in gait parameters between THR performed with standard femoral heads (28-32mm) and large ones (>=36mm).

Aim of the study The aim of this study was to assess potential differences of lower limb biomechanics during gait in patients following total hip replacement surgery depending on femoral head diameter and compare them to the normal gait of healthy volunteers. As a secondary outcome authors wanted to inspect correlation between gait parameters and patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

* BMI <35
* Ability to walk for 10 meters
* 60-80 years of age
* Bilateral THR

Exclusion Criteria:

* Revision surgeries before and after THR
* Any other lower limbs surgeries
* Secondary OA
* Neurological disorders
* Cardiac disorders
* Severly impaired balance
* Severe dizziness

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Time of swing phase | at least 3,5 years after surgery
  Change from baseline part of swing phase time during gait, measured in percentage
Time of stance phase | at least 3,5 years after surgery
  Change from baseline part of stance phase time during gait, measured in percentage
Time of double-stance phase | at least 3,5 years after surgery
  Change from baseline part of double-stance phase time during gait, measured in percentage
Stride length | at least 3,5 years after surgery
  Change from baseline length of stride during gait, measured in meters
Cadence | at least 3,5 years after surgery
  Change from baseline number of strides per minute of walking
Mean gait velocity | at least 3,5 years after surgery
  Change from baseline mean values of gait speed, measured in meters per second
Range of maximal hip extension for both limbs during ending part of mid-stance phase | at least 3,5 years after surgery
  Change from baseline range of maximal hip extension for both limbs during ending part of mid-stance phase, measured in degrees
Range of pelvic drop in frontal plane on the opposite site of the bearing limb | at least 3,5 years after surgery
  Change from baseline range of pelvic drop in frontal plane on the opposite site of the bearing limb, measured in degrees

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz M. Maciąg, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: SAP
Time Frame: The datasets used and/or analyzed during the current study will be available from the corresponding author on reasonable request.
Access Criteria: The datasets used and/or analyzed during the current study will be available from the corresponding author on reasonable request.